CLINICAL TRIAL: NCT00298363
Title: A Phase 2, Double-Blind, Multi-center, Randomized Study Comparing Tenofovir Disoproxil Fumarate, Emtricitabine Plus Tenofovir Disoproxil Fumarate, and Entecavir in the Treatment of Chronic Hepatitis B Subjects With Decompensated Liver Disease and in the Prevention of Hepatitis B Recurrence Post-Transplantation
Brief Title: Study Comparing Tenofovir Disoproxil Fumarate (TDF), Emtricitabine (FTC)/TDF, and Entecavir (ETV) in the Treatment of Chronic HBV in Subjects With Decompensated Liver Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-174-0108
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis; Hepatitis B virus; Tenofovir
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis; Hepatitis B | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tenofovir DF (Experimental): TDF 300 mg + FTC/TDF placebo + ETV placebo once daily (QD)
  Interventions: Drug: Tenofovir disoproxil fumarate (tenofovir DF; TDF); Drug: FTC/TDF placebo; Drug: ETV placebo
- FTC/TDF (Experimental): FTC 200 mg/TDF 300 mg + TDF placebo + ETV placebo QD
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF); Drug: TDF placebo; Drug: ETV placebo
- Entecavir (Experimental): ETV 0.5 mg or 1 mg + TDF placebo + FTC/TDF placebo QD
  Interventions: Drug: Entecavir (ETV); Drug: TDF placebo; Drug: FTC/TDF placebo

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate (tenofovir DF; TDF) — 300-mg tablet QD
  Other Names: Viread
  Arms: Tenofovir DF
Drug: Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) — FTC 200 mg/TDF 300 mg fixed-dose combination (FDC) tablet QD
  Other Names: Truvada
  Arms: FTC/TDF
Drug: Entecavir (ETV) — 0.5-mg or 1-mg tablet QD
  Other Names: Baraclude
  Arms: Entecavir
Drug: TDF placebo — Placebo to match TDF QD
  Arms: Entecavir; FTC/TDF
Drug: FTC/TDF placebo — Placebo to match FTC/TDF QD
  Arms: Entecavir; Tenofovir DF
Drug: ETV placebo — Placebo to match ETV QD
  Arms: FTC/TDF; Tenofovir DF

SUMMARY:
This study was designed to evaluate and compare the safety and tolerability of tenofovir disoproxil fumarate (TDF), emtricitabine (FTC)/TDF, and entecavir (ETV) in the treatment of hepatitis B patients with decompensated liver disease. Safety was assessed by evaluating adverse events (AEs) and laboratory abnormalities. Efficacy was assessed by evaluating reductions in Child-Pugh-Turcotte (CPT) and Model for End Stage Liver Disease (MELD) scores, reductions in hepatitis B virus (HBV) deoxyribonucleic acid (DNA), changes in liver enzymes, development of drug-resistant mutations, and generation of antibody to virus.

A maximum randomized treatment duration of 168 weeks was planned. Since subjects with decompensated liver disease were enrolled into this study, it was necessary to provide early intervention strategies if profound viral suppression was not expeditiously achieved. For this reason, subjects with a decrease in plasma HBV DNA from baseline of < 2 log_10 copies/mL and plasma HBV DNA > 10,000 copies/mL (or plasma HBV DNA > 1,000 copies/mL for subjects who entered the study with HBV DNA < 10,000 copies/mL) at Week 8 had the option to start open-label FTC/TDF and continue in the study. Subjects with a virologic breakthrough or who had plasma HBV DNA levels remaining > 400 copies/mL (confirmed) at or after 24 weeks of treatment could have been unblinded at the investigator's discretion for selection of alternative anti-HBV therapy that may have included open-label FTC/TDF. If study drug was permanently discontinued, immediate initiation of another anti-HBV regimen was strongly recommended.

ELIGIBILITY:
Inclusion Criteria:

A participant was required to meet all of the following inclusion criteria to be eligible for participation in the study:

* Chronic Hepatitis B infection
* 18 through 69 years of age, inclusive
* HBV DNA ≥ 1000 copies/mL
* Decompensated liver disease with all of the following:

  * CPT score of 7-12 (inclusive) OR history of CPT score ≥ 7 and any CPT at screen ≤ 12
  * Serum alanine aminotransferase (ALT) < 10 x the upper limit of the normal range (ULN)
  * Hemoglobin ≥ 7.5 g/dL
  * Total white blood cell (WBC) count ≥ 1,500/mm^3
  * Platelet count ≥ 30,000/mm^3
* Alpha-fetoprotein ≤ 20 ng/mL and ultrasound or other imaging with no evidence of hepatocellular carcinoma (HCC), or alpha-fetoprotein of 21-50 ng/mL and computed tomography (CT)/magnetic resonance imaging (MRI) scan with no evidence of HCC, within 6 months of screening
* Calculated creatinine clearance ≥ 50 mL/min
* Negative human immunodeficiency virus (HIV), hepatitis C virus (HCV), and hepatitis D virus (HDV) serologies
* Less than 24 months of total prior adefovir dipivoxil exposure
* Willing and able to provide written informed consent

Exclusion Criteria:

A participant who met any of the following exclusion criteria could not be enrolled in the study:

* Pregnant women, women who were breastfeeding or who believed they may have wished to become pregnant during the course of the study
* Males and females of reproductive potential who were unwilling to use an effective method of contraception during the study
* Prior use of TDF or ETV
* History of variceal bleeding, hepatorenal syndrome, Grade 3 or 4 hepatic encephalopathy, or spontaneous bacterial peritonitis within 60 days of screening
* Grade 2 hepatic encephalopathy at screening
* History of solid organ or bone marrow transplant
* Current use of hepatotoxic drugs, nephrotoxic drugs, or drugs that interfere with renal tubular secretion
* Current therapy with immunomodulators (eg, corticosteroids, interleukin-2, etc.) or investigational drugs
* Diagnosis of proximal tubulopathy
* Use of investigational agent within 30 days prior to screening
* Known hypersensitivity to TDF, FTC, ETV, or formulation excipients of any of the study drug products

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (38):
- United States (9):
  - Pfleger Liver Institute, Los Angeles, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of Miami, Center for Liver Diseases, Miami, Florida
  - Rush Presbyterian - St. Luke's Medical Center, Chicago, Illinois
  - Henry Ford Hospital and Health System, Detroit, Michigan
  - Mt. Sinai School of Medicine/ Mt. Sinai Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Metropolitan Research, Fairfax, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (4):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - The Gordon & Leslie Diamond Centre, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
- Hopital Conception, Marseille, France
- Germany (3):
  - Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie, Berlin
  - Universitat Heidelberg, Heidelberg
  - Johannes Gutenberg-Universitat, Mainz
- General Hospital of Athens "Ippokratio", Athens, Greece
- Italy (2):
  - Universita de Padova, Padua
  - Policlinico Universitario, Udine
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny im Dluskeigo, Bialystok
  - Wojewodzki Szpital Obserwacy, Bydgoszcz
  - Wojewodzki Szpital Zakazny, Warsaw
- Singapore (4):
  - National University Hospital Dept. of Gastroenterology & Hepatology, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- Spain (5):
  - Hospital General Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona (HCPB), Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario y Politecnico la Fe, Valencia
- Taiwan (4):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaoshiung Hsien
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Taipei
- Turkey (Türkiye) (2):
  - Marmara Universitesi School of Medicine, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir

REFERENCES:
- [Result] Liaw YF, Sheen IS, Lee CM, Akarca US, Papatheodoridis GV, Suet-Hing Wong F, Chang TT, Horban A, Wang C, Kwan P, Buti M, Prieto M, Berg T, Kitrinos K, Peschell K, Mondou E, Frederick D, Rousseau F, Schiff ER. Tenofovir disoproxil fumarate (TDF), emtricitabine/TDF, and entecavir in patients with decompensated chronic hepatitis B liver disease. Hepatology. 2011 Jan;53(1):62-72. doi: 10.1002/hep.23952. Epub 2010 Oct 27. PMID 21254162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 112 participants randomized, 43 were in Taiwan or Singapore, 43 were in Europe (Turkey, Spain, Germany, Greece, Poland, Italy, or France), and 26 were in the US or Canada. The first participant was screened on 04 April 2006, and the last participant was randomized on 03 January 2008. Last participant observation date was 12 April 2011.
Pre-assignment Details: 196 participants screened; 112 randomized and treated (full analysis set; randomized analysis set). Subjects without adequate decrease in HBV DNA at Week 8 could start open-label FTC/TDF. Subjects with virologic breakthrough or HBV DNA levels > 400 copies/mL at ≥ 24 weeks could have received other therapy that may have included open-label FTC/TDF.
Groups:
- Tenofovir DF: Participants in this group were randomized to receive double-blind (DB) TDF 300 mg + FTC)/TDF placebo + ETV placebo at baseline, and may have been unblinded (due to either lack of adequate decrease of HBV DNA or virologic breakthrough) and switched to open-label (OL) FTC/TDF (this study enrolled participants with decompensated liver disease, and early intervention strategies were provided if profound viral suppression was not achieved quickly).
- FTC/TDF: Participants in this group were randomized to receive DB FTC 200 mg/TDF 300 mg + TDF placebo + ETV placebo at baseline, and may have been unblinded (due to either lack of adequate decrease of HBV DNA or virologic breakthrough) and switched to OL FTC/TDF.
- Entecavir: Participants in this group were randomized to receive DB ETV 0.5 mg or 1 mg + TDF placebo + FTC/TDF placebo at baseline, and may have been unblinded (due to either lack of adequate decrease of HBV DNA or virologic breakthrough) and switched to OL FTC/TDF.
Period: Overall Study
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir
Started | 45 | 45 | 22
Completed | 28 (22 completed while taking DB TDF; 6 completed following switch from DB TDF to OL FTC/TDF.) | 37 (34 completed while taking DB FTC/TDF; 3 completed following switch from DB TDF to OL FTC/TDF.) | 16 (13 completed while taking DB ETV; 3 completed following switch from DB ETV to OL FTC/TDF.)
Not Completed | 17 | 8 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 4 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 3
Not completed — Adverse Event | 5 | 2 | 2
Not completed — Lack of Efficacy | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tenofovir DF: Participants in this group were randomized to receive TDF 300 mg + FTC/TDF placebo + ETV placebo at baseline
- FTC/TDF: Participants in this group were randomized to receive FTC 200 mg/TDF 300 mg + TDF placebo + ETV placebo at baseline
- Entecavir: Participants in this group were randomized to receive ETV 0.5 mg or 1 mg + TDF placebo + FTC/TDF placebo at baseline
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Total
Number analyzed (Participants) | 45 | 45 | 22 | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (8.8) | 49 (10.1) | 52 (12.0) | 51 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 18
  Male | 37 | 40 | 17 | 94
Region of Enrollment [Number; unit: participants]
  France | 0 | 0 | 1 | 1
  United States | 10 | 2 | 2 | 14
  Taiwan | 13 | 16 | 9 | 38
  Greece | 4 | 1 | 1 | 6
  Canada | 4 | 7 | 1 | 12
  Poland | 2 | 2 | 2 | 6
  Spain | 2 | 6 | 2 | 10
  Singapore | 1 | 3 | 1 | 5
  Turkey | 4 | 6 | 2 | 12
  Germany | 4 | 1 | 1 | 6
  Italy | 1 | 1 | 0 | 2
Race [Number; unit: participants]
  Asian | 23 | 24 | 13 | 60
  Black | 1 | 1 | 0 | 2
  Other | 2 | 0 | 1 | 3
  White | 19 | 20 | 8 | 47
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 39 | 39 | 21 | 99
  Not Permitted | 4 | 5 | 1 | 10
Weight [Mean (Standard Deviation); unit: kg] | 78.1 (17.02) | 74.4 (15.41) | 77.3 (16.64) | 76.5 (16.26)
Height [Mean (Standard Deviation); unit: cm] | 168.3 (7.98) | 168.4 (8.47) | 167.1 (8.39) | 168.1 (8.20)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (5.67) | 26.2 (5.07) | 27.6 (5.27) | 27.0 (5.35)

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Tolerability Failure
Description: Tolerability failure was defined as permanent discontinuation of study drug due to a treatment-emergent adverse event (AE), including any subject who temporarily discontinued study drug due to an AE and did not restart. Results are expressed as proportions of participants who experience tolerability failure using the Kaplan-Meier (KM) method of estimation.
Time Frame: Baseline to Week 168
Population: Full analysis set (all randomized subjects who received at least one dose of study drug)
Measure: Number (95% Confidence Interval); unit: percent probability (KM estimate)
Groups:
- TDF or FTC/TDF: Participants in this group include all participants who received TDF or FTC/TDF during the study.
Arm/Group | Tenofovir DF | FTC/TDF | TDF or FTC/TDF | Entecavir
Number analyzed (Participants) | 45 | 45 | 90 | 22
percent probability (KM estimate) | 18 [5.8 to 30.6] | 4 [0.0 to 10.4] | 11 [4.1 to 17.7] | 14 [0.0 to 29.5]

2. Secondary Outcome: Median Time-averaged Change (DAVG) in Plasma Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels at 48 Weeks Relative to Baseline
Description: Change from baseline was evaluated by subtracting baseline HBV DNA log_10 copies/mL from Week 48 HBV DNA log_10 copies/mL. DAVG is defined as the area of the trapezoid under the response-time curve divided by time to the last available evaluation of the patient minus the baseline value.
Time Frame: Baseline to 48 weeks
Population: Participants with HBV DNA measurements at Week 48 were included in this analysis.
Measure: Median (Inter-Quartile Range); unit: log_10 copies/mL
Groups:
- Overall: Participants in this group includes all participants from TDF, FTC/TDF, and ETV groups
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 36 | 38 | 18 | 92
log_10 copies/mL | -2.93 [-3.84 to -2.18] | -3.45 [-4.73 to -2.02] | -3.61 [-4.51 to -1.31] | -3.19 [-4.52 to -2.08]

3. Secondary Outcome: Median DAVG in Plasma HBV DNA Levels at 96 Weeks Relative to Baseline
Description: Change from baseline was evaluated by subtracting baseline HBV DNA log_10 copies/mL from Week 96 HBV DNA log_10 copies/mL. DAVG is defined as the area of the trapezoid under the response-time curve divided by time to the last available evaluation of the patient minus the baseline value.
Time Frame: Baseline to 96 weeks
Population: Full analysis set; data collected for participants who underwent liver transplant prior to Week 96 were excluded.
Measure: Median (Inter-Quartile Range); unit: log_10 copies/mL
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 34 | 35 | 16 | 85
log_10 copies/mL | -3.06 [-4.17 to -2.18] | -4.06 [-4.97 to -2.38] | -3.32 [-4.82 to -1.26] | -3.40 [-4.81 to -2.14]

4. Secondary Outcome: Median DAVG in Plasma HBV DNA Levels at 144 Weeks Relative to Baseline
Description: Change from baseline was evaluated by subtracting baseline HBV DNA log_10 copies/mL from Week 144 HBV DNA log_10 copies/mL. DAVG is defined as the area of the trapezoid under the response-time curve divided by time to the last available evaluation of the patient minus the baseline value.
Time Frame: Baseline to 144 weeks
Population: Full analysis set; data collected for participants who underwent liver transplant prior to Week 144 were excluded.
Measure: Median (Inter-Quartile Range); unit: log _10 copies/mL
Groups:
- FTC/TDF: Participants in this group were randomized to receive FTC 200mg/TDF 300 mg + TDF placebo + ETV placebo at baseline
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 28 | 34 | 15 | 77
log _10 copies/mL | -3.07 [-4.36 to -2.00] | -3.82 [-4.99 to -2.06] | -3.76 [-5.00 to -1.33] | -3.49 [-4.91 to -2.05]

5. Secondary Outcome: Median DAVG in Plasma HBV DNA Levels at 168 Weeks Relative to Baseline
Description: Change from baseline was evaluated by subtracting baseline HBV DNA log_10 copies/mL from Week 168 HBV DNA log_10 copies/mL. DAVG is defined as the area of the trapezoid under the response-time curve divided by time to the last available evaluation of the patient minus the baseline value.
Time Frame: Baseline to 168 weeks
Population: Full analysis set; data collected for participants who underwent liver transplant prior to Week 168 were excluded.
Measure: Median (Inter-Quartile Range); unit: log_10 copies/mL
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 26 | 31 | 15 | 72
log_10 copies/mL | -3.16 [-4.57 to -1.97] | -4.06 [-5.15 to -2.42] | -3.77 [-5.02 to -1.33] | -3.66 [-4.99 to -2.10]

6. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 400 Copies/mL at Week 48
Description: The percentage of participants with plasma HBV DNA < 400 copies/mL at Week 48 was summarized.
Time Frame: Week 48
Population: Full analysis set; noncompleters/switch = failure analysis (participants who did not complete treatment or changed from double-blind to open-label treatment up to the time point were considered as failing to meet efficacy response criteria [defined as not achieving viral suppression of < 400 copies/mL]).
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 44 | 41 | 22 | 107
percentage of participants | 70.5 | 87.8 | 72.7 | 77.6

7. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 400 Copies/mL at Week 96
Description: The percentage of participants with plasma HBV DNA < 400 copies/mL at Week 96 was summarized.
Time Frame: Week 96
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 44 | 39 | 21 | 104
percentage of participants | 59.1 | 79.5 | 57.1 | 66.3

8. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 400 Copies/mL at Week 144
Description: The percentage of participants with plasma HBV DNA < 400 copies/mL at Week 144 was summarized.
Time Frame: Week 144
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 44 | 40 | 21 | 105
percentage of participants | 50.0 | 77.5 | 52.4 | 61.0

9. Secondary Outcome: Percentage of Participants With Plasma HBV DNA < 400 Copies/mL at Week 168
Description: The percentage of participants with plasma HBV DNA < 400 copies/mL at Week 168 was summarized.
Time Frame: Week 168
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 42 | 37 | 21 | 100
percentage of participants | 50.0 | 75.7 | 52.4 | 60.0

10. Secondary Outcome: Percentage of Participants With Normalized Alanine Aminotransferase (ALT) (for Subjects With Elevated ALT at Baseline) at Week 48
Description: Normalized ALT is defined as having a baseline ALT value > the upper limit of the normal range (ULN), and a decrease in ALT value to ≤ ULN at the given time point.
Time Frame: Baseline to Week 48
Population: Biochemically evaluable analysis set (subjects in full analysis set with abnormal baseline alanine aminotransferase [ALT] values); noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 26 | 25 | 17 | 68
percentage of participants | 46.2 | 64.0 | 41.2 | 51.5

11. Secondary Outcome: Percentage of Participants With Normalized ALT (for Subjects With Elevated ALT at Baseline) at Week 96
Description: Normalized ALT is defined as having a baseline ALT value > ULN, and a decrease in ALT value to ≤ ULN at the given time point.
Time Frame: Baseline to Week 96
Population: Biochemically evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 26 | 24 | 16 | 66
percentage of participants | 50.0 | 58.3 | 31.3 | 48.5

12. Secondary Outcome: Percentage of Participants With Normalized ALT (for Subjects With Elevated ALT at Baseline) at Week 144
Description: as for outcome 11
Time Frame: Baseline to Week 144
Population: Biochemically evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 26 | 25 | 16 | 67
percentage of participants | 34.6 | 64.0 | 37.5 | 46.3

13. Secondary Outcome: Percentage of Participants With Normalized ALT (for Subjects With Elevated ALT at Baseline) at Week 168
Description: as for outcome 11
Time Frame: Baseline to Week 168
Population: Biochemically evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 24 | 25 | 16 | 65
percentage of participants | 29.2 | 60.0 | 37.5 | 43.1

14. Secondary Outcome: Percentage of Participants With an Increase in Child-Pugh Turcotte (CPT) Score of ≥ 2 Points at Weeks 48
Description: CPT scores, widely used to grade the severity of cirrhosis and to determine the need for liver transplantation, are calculated based on a combination of laboratory values and clinical features. CPT scores can range from 5 to 15, with higher scores indicating a greater severity of disease.
Time Frame: Baseline to Week 48
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 43 | 38 | 22 | 103
percentage of participants | 0.0 | 2.6 | 0.0 | 1.0

15. Secondary Outcome: Percentage of Participants With an Increase in CPT Score of ≥ 2 Points at Week 96
Description: as for outcome 14
Time Frame: Baseline to Week 96
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 43 | 38 | 20 | 101
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

16. Secondary Outcome: Percentage of Participants With an Increase in CPT Score of ≥ 2 Points at Week 144
Description: as for outcome 14
Time Frame: Baseline to Week 144
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 43 | 40 | 21 | 104
percentage of participants | 0.0 | 2.5 | 0.0 | 1.0

17. Secondary Outcome: Percentage of Participants With an Increase in CPT Score of ≥ 2 Points at Week 168
Description: as for outcome 14
Time Frame: Baseline to Week 168
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 41 | 36 | 21 | 98
percentage of participants | 2.4 | 0.0 | 0.0 | 1.0

18. Secondary Outcome: Percentage of Participants With a Decrease in CPT Score of ≥ 2 Points From Baseline at Week 48
Description: as for outcome 14
Time Frame: Baseline to Week 48
Population: CPT evaluable analysis set (subjects with CPT scores ≥ 7 at baseline; because the minimum CPT score was 5, only these subjects were evaluable for analyses of ≥ 2-point decrease in CPT score); noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 27 | 25 | 12 | 64
percentage of participants | 25.9 | 48.0 | 41.7 | 37.5

19. Secondary Outcome: Percentage of Participants With a Decrease in CPT Score of ≥ 2 Points From Baseline at Week 96
Description: as for outcome 14
Time Frame: Baseline to Week 96
Population: CPT evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 26 | 25 | 10 | 61
percentage of participants | 23.1 | 52.0 | 50.0 | 39.3

20. Secondary Outcome: Percentage of Participants With a Decrease in CPT Score of ≥ 2 Points From Baseline at Week 144
Description: as for outcome 14
Time Frame: Baseline to Week 144
Population: CPT evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 27 | 27 | 11 | 65
percentage of participants | 25.9 | 51.9 | 45.5 | 40.0

21. Secondary Outcome: Percentage of Participants With a Decrease in CPT Score of ≥ 2 Points From Baseline at Week 168
Description: as for outcome 14
Time Frame: Baseline to Week 168
Population: CPT evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 25 | 24 | 11 | 60
percentage of participants | 24.0 | 45.8 | 45.5 | 36.7

22. Secondary Outcome: Median Change in Model for End-Stage Liver Disease (MELD) Score From Baseline at Week 48
Description: MELD scores, used to assess prognosis and suitability for transplant, are calculated based on laboratory values only and can range from 6 to 40, with higher scores indicating greater disease severity.
Time Frame: Baseline to Week 48
Population: Subjects in the full analysis set with an available score at the visit
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 35 | 35 | 19 | 89
units on a scale | -2.0 [-3.0 to 0.0] | -2.0 [-4.0 to 0.0] | -2.0 [-4.0 to -1.0] | -2.0 [-3.0 to 0.0]

23. Secondary Outcome: Median Change in MELD Score From Baseline at Week 96
Description: as for outcome 22
Time Frame: Baseline to Week 96
Population: Subjects in the full analysis set with an available score at the visit
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 33 | 33 | 15 | 81
units on a scale | -2.0 [-3.0 to 1.0] | -3.0 [-4.0 to 0.0] | -3.0 [-4.0 to -1.0] | -2.0 [-4.0 to 0.0]

24. Secondary Outcome: Median Change in MELD Score From Baseline at Week 144
Description: as for outcome 22
Time Frame: Baseline to Week 144
Population: Subjects in the full analysis set with an available score at the visit
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 28 | 34 | 15 | 77
units on a scale | -2.0 [-3.5 to -0.5] | -1.5 [-6.0 to 0.0] | -2.0 [-5.0 to -1.0] | -2.0 [-4.0 to 0.0]

25. Secondary Outcome: Median Change in MELD Score From Baseline at Week 168
Description: as for outcome 22
Time Frame: Baseline to Week 168
Population: Subjects in the full analysis set with an available score at the visit
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 25 | 30 | 15 | 70
units on a scale | -2.0 [-4.0 to -1.0] | -2.0 [-4.0 to 0.0] | -2.0 [-5.0 to 0.0] | -2.0 [-4.0 to 0.0]

26. Secondary Outcome: Percentage of Participants With Hepatitis B Early Antigen (HBeAg) Loss and HBeAg Seroconversion at Week 48 (for Participants Who Were HBeAg Positive at Baseline)
Description: Loss of HBeAg was defined as change of detectable HBeAg from positive to negative. HBeAg seroconversion was defined as change of detectable antibody to HBeAg from negative to positive.
Time Frame: Baseline to Week 48
Population: Serologically evaluable analysis set (subjects in full analysis set with positive hepatitis B early antigen [HBeAg] at baseline); noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 14 | 15 | 7 | 36
percentage of participants
  HBeAg Loss | 21.4 | 26.7 | 0.0 | 19.4
  HBeAg Seroconversion | 21.4 | 13.3 | 0.0 | 13.9

27. Secondary Outcome: Percentage of Participants With HBeAg Loss and HBeAg Seroconversion at Week 96 (for Participants Who Were HBeAg Positive at Baseline)
Description: as for outcome 26
Time Frame: Baseline to Week 96
Population: Serologically evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 14 | 15 | 6 | 35
percentage of participants
  HBeAg Loss | 14.3 | 33.3 | 0.0 | 20.0
  HBeAg Seroconversion | 14.3 | 13.3 | 0.0 | 11.4

28. Secondary Outcome: Percentage of Participants With HBeAg Loss and HBeAg Seroconversion at Week 144 (for Participants Who Were HBeAg Positive at Baseline)
Description: as for outcome 26
Time Frame: Baseline to Week 144
Population: Serologically evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 14 | 15 | 6 | 35
percentage of participants
  HBeAg Loss | 14.3 | 33.3 | 16.7 | 22.9
  HBeAg Seroconversion | 14.3 | 13.3 | 0.0 | 11.4

29. Secondary Outcome: Percentage of Participants With HBeAg Loss and HBeAg Seroconversion at Week 168 (for Participants Who Were HBeAg Positive at Baseline)
Description: as for outcome 26
Time Frame: Baseline to Week 168
Population: Serologically evaluable analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 13 | 14 | 6 | 33
percentage of participants
  HBeAg Loss | 23.1 | 35.7 | 16.7 | 27.3
  HBeAg Seroconversion | 23.1 | 21.4 | 0.0 | 18.2

30. Secondary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Loss and HBsAg Seroconversion at Week 48
Description: Loss of HBsAg was defined as change of detectable HBsAg from positive to negative. HBsAg seroconversion was defined as change of detectable antibody to HBsAg from negative to positive.
Time Frame: Baseline to Week 48
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 43 | 41 | 22 | 106
percentage of participants
  HBsAg Loss | 0.0 | 0.0 | 0.0 | 0.0
  HBsAg Seroconversion | 0.0 | 0.0 | 0.0 | 0.0

31. Other Pre Specified Outcome: Percentage of Participants With Only Baseline Adefovir Dipivoxil Resistance (ADV-R) Mutations Achieving HBV DNA < 400 Copies/mL by 168 Weeks
Description: ADV resistance mutations are defined as the presence of the rtA181T/V HBV gene mutation and/or the rtN236T HBV gene mutation.
Time Frame: Baseline to Week 168
Population: Participants in the full analysis set with ADV resistance mutation at baseline were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir
Number analyzed (Participants) | 1 | 1 | 0
percentage of participants | 100 | 100 |

32. Other Pre Specified Outcome: Percentage of Participants With Only Baseline Lamivudine-resistance (LAM-R) Mutations Achieving HBV DNA < 400 Copies/mL by 168 Weeks
Description: LAM resistance mutations are defined as the presence of the rtM204V/I HBV gene mutation with or without the rtL180M HBV gene mutation.
Time Frame: Baseline to Week 168
Population: Patients in the full analysis set with LAM resistance mutation at baseline were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir
Number analyzed (Participants) | 5 | 8 | 3
percentage of participants | 100 | 100 | 100

33. Other Pre Specified Outcome: Percentage of Participants With Baseline ADV-R + LAM-R Mutations Achieving HBV DNA < 400 Copies/mL by 168 Weeks
Description: ADV resistance mutation + LAM resistance mutations are defined as the presence of the rtA181T/V HBV gene mutation and/or the rtN236T HBV gene mutation, and the rtM204V/I HBV gene mutation with or without the rtL180M HBV gene mutation.
Time Frame: Baseline to Week 168
Population: Participants in the full analysis set with both ADV and LAM resistance mutations at baseline were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir
Number analyzed (Participants) | 2 | 0 | 0
percentage of participants | 50 |  |

34. Primary Outcome: Percent Probability of a Confirmed Increase in Serum Creatinine of ≥ 0.5 mg/dL From Baseline or a Confirmed Serum Phosphorus Level < 2.0 mg/dL
Description: Results are expressed as proportions of participants who experience a confirmed increase in serum creatinine of ≥ 0.5 mg/dL from baseline or a confirmed serum phosphorus level < 2.0 mg/dL using the KM method of estimation.
Time Frame: Baseline to Week 168
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percent probability (KM estimate)
Arm/Group | Tenofovir DF | FTC/TDF | TDF or FTC/TDF | Entecavir
Number analyzed (Participants) | 45 | 45 | 90 | 22
percent probability (KM estimate) | 15 [3.9 to 25.9] | 14 [3.6 to 24.4] | 14 [6.8 to 22.0] | 10 [0.0 to 22.8]

35. Secondary Outcome: Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 96
Description: as for outcome 30
Time Frame: Baseline to Week 96
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 44 | 39 | 21 | 104
percentage of participants
  HBsAg Loss | 0.0 | 0.0 | 0.0 | 0.0
  HBsAg Seroconversion | 0.0 | 0.0 | 0.0 | 0.0

36. Secondary Outcome: Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 144
Description: as for outcome 30
Time Frame: Baseline to Week 144
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 43 | 38 | 21 | 102
percentage of participants
  HBsAg Loss | 0.0 | 0.0 | 0.0 | 0.0
  HBsAg Seroconversion | 0.0 | 0.0 | 0.0 | 0.0

37. Secondary Outcome: Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 168
Description: as for outcome 30
Time Frame: Baseline to Week 168
Population: Full analysis set; noncompleters/switch = failure
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 41 | 36 | 21 | 98
percentage of participants
  HBsAg Loss | 0.0 | 0.0 | 0.0 | 0.0
  HBsAg Seroconversion | 0.0 | 0.0 | 0.0 | 0.0

38. Secondary Outcome: In the Subset of Participants Undergoing Liver Transplantation, Time to Recurrence of Hepatitis B, Defined as 2 Consecutive Plasma HBV DNA Concentrations ≥ 400 Copies/mL or 2 Consecutive HBsAg(+) Results
Time Frame: Baseline to Week 168
Population: Liver transplantation analysis set
Measure: Number; unit: Days
Arm/Group | Tenofovir DF | FTC/TDF | Entecavir | Overall
Number analyzed (Participants) | 3 | 7 | 1 | 11
Days | NA — No participant in this category experienced Hepatitis B Recurrence. | NA — No participant in this category experienced Hepatitis B Recurrence. | NA — No participant in this category experienced Hepatitis B Recurrence. | NA — No participant in this category experienced Hepatitis B Recurrence.

ADVERSE EVENTS:
Groups:
- Double Blind TDF: Participants in this group were randomized to receive TDF 300 mg + FTC/TDF placebo + ETV placebo
- Double Blind FTC/TDF: Participants in this group were randomized to receive FTC 200 mg/TDF 300 mg + TDF placebo + ETV placebo
- Double Blind ETV: Participants in this group were randomized to receive ETV 0.5 mg or 1 mg + TDF placebo + FTC/TDF placebo
- Open Label FTC/TDF: Participants in this group were randomized to receive TDF, FTC/TDF, or ETV at the beginning of the study, but switched to open label FTC/TDF during the study.
- All TDF: Participants in this group received a TDF-containing treatment (all double-blind TDF, FTC/TDF, or open-label FTC/TDF) during the study.
Arm/Group | Double Blind TDF | Double Blind FTC/TDF | Double Blind ETV | Open Label FTC/TDF | All TDF
Serious Adverse Events (participants affected / at risk) | 21/45 | 25/45 | 11/22 | 4/12 | 50/93
Other Adverse Events (participants affected / at risk) | 41/45 | 44/45 | 20/22 | 9/12 | 89/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind TDF (N=45) | Double Blind FTC/TDF (N=45) | Double Blind ETV (N=22) | Open Label FTC/TDF (N=12) | All TDF (N=93)
Ascites (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 7
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 4
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 5 | 2 | 0 | 7
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 3
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Porcelain gallbladder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 2 | 3 | 0 | 0 | 5
Sepsis (Infections and infestations) | 1 | 3 | 0 | 0 | 4
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Scrotal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3 | 2 | 1 | 12
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 3 | 1 | 2 | 0 | 4
Encephalopathy (Nervous system disorders) | 1 | 2 | 0 | 0 | 3
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Cerebrospinal fluid rhinorrhoea (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Device failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Traumatic spinal cord compression (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1
Generalized oedema (General disorders) | 1 | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal aneurysm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Liver transplant rejection (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Mental status change (Psychiatric disorders) | 2 | 0 | 0 | 0 | 2
Schizophreniform disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind TDF (N=45) | Double Blind FTC/TDF (N=45) | Double Blind ETV (N=22) | Open Label FTC/TDF (N=12) | All TDF (N=93)
Abdominal pain upper (Gastrointestinal disorders) | 9 | 7 | 2 | 2 | 18
Ascites (Gastrointestinal disorders) | 8 | 4 | 6 | 1 | 13
Abdominal pain (Gastrointestinal disorders) | 6 | 4 | 3 | 1 | 11
Nausea (Gastrointestinal disorders) | 9 | 3 | 1 | 0 | 12
Abdominal distension (Gastrointestinal disorders) | 5 | 4 | 2 | 1 | 10
Vomiting (Gastrointestinal disorders) | 6 | 2 | 2 | 1 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 6 | 1 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 5 | 1 | 5
Constipation (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 5
Inguinal hernia (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 5
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 5 | 7 | 1 | 0 | 12
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 2 | 2 | 9
Urinary tract infection (Infections and infestations) | 4 | 2 | 1 | 1 | 7
Bronchitis (Infections and infestations) | 3 | 1 | 2 | 1 | 5
Peritonitis bacterial (Infections and infestations) | 2 | 3 | 0 | 0 | 5
Sepsis (Infections and infestations) | 2 | 3 | 0 | 0 | 5
Influenza (Infections and infestations) | 1 | 2 | 0 | 1 | 4
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 5 | 2 | 0 | 7
Cholelithiasis (Hepatobiliary disorders) | 2 | 4 | 0 | 0 | 6
Jaundice (Hepatobiliary disorders) | 1 | 3 | 1 | 0 | 4
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1 | 0 | 2 | 4
Portal hypertension (Hepatobiliary disorders) | 2 | 1 | 0 | 1 | 4
Hepatomegaly (Hepatobiliary disorders) | 2 | 0 | 0 | 1 | 3
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 8 | 3 | 5 | 0 | 11
Pyrexia (General disorders) | 6 | 5 | 4 | 0 | 11
Asthenia (General disorders) | 5 | 2 | 2 | 0 | 7
Fatigue (General disorders) | 2 | 2 | 2 | 0 | 4
Chest pain (General disorders) | 1 | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2 | 0 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 4 | 3 | 5 | 1 | 8
Dizziness (Nervous system disorders) | 6 | 3 | 0 | 0 | 9
Hepatic encephalopathy (Nervous system disorders) | 5 | 2 | 3 | 0 | 7
Encephalopathy (Nervous system disorders) | 3 | 3 | 0 | 0 | 6
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 6 | 2 | 0 | 13
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 1 | 1 | 10
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 2 | 2 | 1 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 3
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 9 | 4 | 4 | 1 | 14
Depression (Psychiatric disorders) | 2 | 1 | 1 | 1 | 4
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 2 | 8
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 3
Chronic obstructrive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 2 | 0 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 0 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Cardiac murmur (Investigations) | 2 | 1 | 0 | 1 | 4
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3 | 2 | 1 | 12
Renal failure (Renal and urinary disorders) | 2 | 0 | 1 | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 2
Calculus Ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 5 | 0 | 1 | 7
Hypotension (Vascular disorders) | 4 | 0 | 0 | 0 | 4
Gynaecomastia (Reproductive system and breast disorders) | 2 | 3 | 1 | 1 | 6
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 2 | 1 | 3
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 2
Creatinine renal clearance increased (Investigations) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years